CLINICAL TRIAL: NCT00975325
Title: Characterisation of Relative Bioavailability and Assessment of Bioequivalence of Two Generic Yohimbine Formulations in Comparison With a Marketed Reference Product - an Open, Randomised, Single Dose, 3-period Change-over Study
Brief Title: Bioequivalence Study Comparing Two Test Products With One Reference Product, All Containing 5 mg Yohimbine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Ritter GmbH & Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YOH-BE-2009; EudraCT No.2009-013122-16
Record Dates: First submitted 2009-09-08; First posted 2009-09-11 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Erectile Dysfunction
Keywords: Bioequivalency
MeSH Terms: conditions — Erectile Dysfunction | interventions — Yohimbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yohimbine, Yohimbine "Spiegel" (Active Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine Yocon-Glenwood (Active Comparator)
  Interventions: Drug: Yohimbine

INTERVENTIONS:
Drug: Yohimbine — yohimbine 5 mg, one tablet, single dose only
  Arms: Yohimbine, Yohimbine "Spiegel"
Drug: Yohimbine — yohimbine 5 mg, one tablet, single dose only
  Arms: Yohimbine Yocon-Glenwood

SUMMARY:
* Type: Bioequivalence study in male healthy volunteers, therapeutical indication (erectile disfunction) not studied
* Products, dosage, and route of administration:

  * Test 1: Yohimbin "Spiegel"® (Desma GmbH, Germany), tablet containing 5 mg yohimbine hydrochloride, oral administration
  * Reference: Yocon-Glenwood® (Glenwood GmbH, Germany), tablet containing 5 mg yohimbine hydrochloride, oral administration
* Duration of treatment:

  2 single-dose administrations of 5 mg yohimbine hydrochloride each under fasting conditions separated by a wash-out period of at least one week i.e. 6 treatment free days between all administrations

DETAILED DESCRIPTION:
Study objectives

Primary Objectives:

* Characterisation of relative bioavailability of Test 1 in comparison to Reference after single dose administration under fasting conditions
* Assessment of bioequivalence of Test 1 vs. Reference after single dose administration under fasting conditions, determined by use of area under the concentration time curve AUC0-tlast and maximal concentration Cmax obtained for yohimbine

Secondary Objective:

* Descriptive characterisation of safety and tolerability of the investigational products in the study population
* Descriptive characterisation of blood pressure and pulse rate around Cmax of the investigational products in the study population

Analytical methodology:

Yohimbine in plasma samples will be analysed by use of a validated HPLC-MS/MS; intended LLOQ for yohimbine is 0.5 ng/ml

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Ethnic origin: Caucasian
* Age: 18 - 55 years, inclusive
* Body-mass index1 (BMI): ≥ 19 kg/m² and ≤ 27 kg/m²
* Good state of health
* Non-smoker or an ex-smoker for a least 1 month
* Written informed consent, after having been informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subjects participating in the study

Exclusion Criteria:

* Safety concerns:

  1. Existing cardiac or haematological diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
  2. Existing hepatic and/or renal diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
  3. Existing gastrointestinal diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
  4. History of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
  5. Pathological ECG (12 standard leads) which might interfere with the safety of the active ingredient
  6. Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
  7. Subjects with severe allergies or multiple drug allergies
  8. Systolic blood pressure <100/>140 mmHg
  9. Diastolic blood pressure <60/>90 mmHg
  10. Pulse rate <45/>110 bpm
  11. Laboratory values out of normal range unless the deviation from normal is judged as not relevant for the study by the investigator
  12. Positive anti-HIV-test, HBs-AG-test or anti-HCV-test
  13. History of glaucoma
* Lack of suitability for the trial 14. Subjects exhibiting extreme genetic polymorphism of CYP 2D6 - "Poor or Ultra-rapid metabolizer" 15. Acute or chronic diseases which could affect absorption or metabolism 16. History of or current drug or alcohol dependence 17. Regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male per day 18. Subjects who are on a diet which could affect the pharmacokinetics of the active ingredient 19. Regular intake of caffeine containing food or beverages of ≥ 500 mg per day 20. Blood donation or other blood loss of more than 400 ml within the last two months prior to individual enrolment of the subject 21. Participation in a clinical trial during the last two months prior to individual enrolment of the subject 22. Regular treatment with any systemically available medication (except continuous usual replacement therapy e.g. L-thyroxine) within two weeks prior to the first administration of the study medication 23. Intake of yohimbine for any reason (e.g. fat burning, weight reduction, muscle improvement, post operative care and/or any therapy for erectile dysfunctions) within two weeks prior to first administration of the study medication 24. Subjects, who report a frequent occurrence of migraine attacks
* Administrative reasons 25. Subjects suspected or known not to follow instructions 26. Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter AUC, Cmax | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- SocraTec R&D GmbH, Erfurt, Germany